CLINICAL TRIAL: NCT04371198
Title: Feasibility of Establishing Patient-Derived Organoids for Rectal Cancer: A Biospecimen Collection Protocol
Brief Title: Patient-Derived Organoids for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00104561
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-10

CONDITIONS: Rectum Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organoid (Experimental)
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Tissue biopsy

SUMMARY:
The purpose of this study is to determine the feasibility of establishing patient-derived organoids from pre-treatment rectal adenocarcinoma biopsies.

ELIGIBILITY:
Inclusion

1. Age ≥18 years old.
2. Able to provide informed consent.
3. Undergoing proctoscopy.

Exclusion

1. Patient not planned to receive neoadjuvant radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czito, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and organoids may be shared with other researchers
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication
Access Criteria: Researchers should request data and/or organoid lines from the principal investigator

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Organoid
Started | 20
Completed | 16
Not Completed | 4
Not completed — inadequate sample | 4

BASELINE CHARACTERISTICS:
Arm/Group | Organoid
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsies That Form Spherical Organoids
Time Frame: Baseline
Population: Participants with sufficient sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Organoid
Number analyzed (Participants) | 16
Participants | 14

ADVERSE EVENTS:
Time Frame: Adverse Event data was not collected.
Description: Adverse Event data was not collected.
Arm/Group | Organoid
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04371198/Prot_SAP_000.pdf